CLINICAL TRIAL: NCT01634009
Title: Efficacy of Ready to Use Therapeutic Food Using Soy Protein Isolate in Under-5 Children With Severe Acute Malnutrition in Bangladesh
Brief Title: Soy-Ready to Use Therapeutic Food (RUTF) in Severely Malnourished Children
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: International Centre for Diarrhoeal Disease Research, Bangladesh (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: PR-09038
Record Dates: First submitted 2012-06-12; First posted 2012-07-06 (Estimated); Last update posted 2017-09-25 (Actual); Status verified 2016-06

CONDITIONS: Severe Acute Malnutrition; Severe Wasting; Community Based Nutritional Management
Keywords: Severe acute malnutrition; Ready to use therapeutic food; Soy protein; Community based management; Efficacy; Management of Children with SAM in Bangladesh
MeSH Terms: conditions — Severe Acute Malnutrition; Cachexia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard RUTF (control) (Active Comparator): Children will receive standard RUTF in this arm and will be considered as control arm
  Interventions: Dietary Supplement: Soy-based RUTF (in double blind design)
- Standard RUTF (No Intervention): Will act as control

INTERVENTIONS:
Dietary Supplement: Soy-based RUTF (in double blind design) — Soy-based RUTF will be given in double blind manner
  Other Names: Soy-based RUTF is the intervention
  Arms: Standard RUTF (control)

SUMMARY:
SAM defined by having weight-for-height (WH) less than - 3 Z score or bi-pedal nutritional edema is an important cause of death in children globally including Bangladesh. The death rate among children hospitalized for SAM is still high. Severe malnutrition in children can be successfully treated by using WHO guidelines with or without minor modification. Since the Community Based Therapeutic Care (CTC)/CMAM approach was developed, the use of RUTF for the treatment of children with SAM has gained ground, and huge amounts of RUTF are used particularly in African countries. RUTFs are an energy-dense lipid paste enriched with vitamins and minerals. The typical composition (ingredient % of weight) of RUTF is whole milk powder 30%; sugar 28%; vegetable oil 15.4%; peanut paste 25%; and mineral vitamin mix 1.6%. Although the CTC model promises treatment of SAM at a considerably lower cost than the previous inpatient model, the cost of RUTF is still considered a significant barrier to universal roll-out of SAM treatment and has made CTC implementation too expensive in many high-need countries.

The single most expensive raw ingredient in RUTF is milk powder, contributing around 50% of raw ingredient cost or between 30-35% of the total cost of the final product. Isolated soy protein has a cost per kg protein that normally is below that of skim or whole milk powder, and can thus reduce the total cost of RUTF. In addition, isolated soy protein (ISP) is a high quality, complete protein that meets the daily protein requirements of growing children and adults. ISP is a highly digestible protein [FAO/WHO, 1991] with an amino acid profile that has been shown to achieve a Protein Digestibility-Corrected Amino Acid Score (PDCAAS) of 1.00, comparable to milk and eggs, and has been shown to maintain nitrogen balance when fed as the sole protein source at minimum recommended intake levels.

To compare the efficacy (weight gain, rate of weight gain and change of lean body mass) of the standard RUTF and an RUTF made from ISP (Soy-RUTF) through a randomized double masked intervention trial 300 SAM children aged 6 to 59 months after completion of their stabilization phase from the Dhaka Hospital of icddr,b Bangladesh will be studied. They will randomly receive standard- or Soy-RUTF as take home and followed up (weekly until achieving -2 WHZ, and thereafter fortnightly until achieving -1 WHZ) at the nutrition follow up unit at the outpatient department of this Dhaka Hospital of icddr,b.

ELIGIBILITY:
Inclusion Criteria:

* children (both boys and girls) with SAM defined by WH < -3 Z score of WHO standard,
* completed acute (stabilization) phase management,
* clinically well,
* no edema and regaining appetite and aged 6 to 60 months will be included. - additional enrollment criteria will be as follows:

  * no signs of concurrent infection,
  * mothers/caregivers agreed to stay in their current address for next 4 months (for tracking the children)

Exclusion Criteria:

* failure to obtain consent from parents or caretakers;
* children without any fixed address;
* children with tuberculosis or any congenital/acquired disorder affecting growth i.e. trisomy-21 or cerebral palsy;
* children on an exclusion diet for the treatment of persistent diarrhea,
* having history of soy, peanut or milk protein allergy.

Ages: 6 Months to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 260 (Actual)
Dates: Start 2012-07; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
To compare the efficacy (rate of weight gain) | 31 December 2014 (up to 3 years)
  By 31st December 2014 we shall be able to complete the enrollment, data analyses and preliminary/draft report writting.

CONTACTS AND LOCATIONS:
Overall Officials: MD IQBAL HOSSAIN, DCH, PhD, Principal Investigator — International Centre for Diarrhoeal Disease Research, Bangladesh
Locations (1):
- Icddr,B, Dhaka, Bangladesh

REFERENCES:
- [Derived] Hossain MI, Huq S, Islam MM, Ahmed T. Acceptability and efficacy of ready-to-use therapeutic food using soy protein isolate in under-5 children suffering from severe acute malnutrition in Bangladesh: a double-blind randomized non-inferiority trial. Eur J Nutr. 2020 Apr;59(3):1149-1161. doi: 10.1007/s00394-019-01975-w. Epub 2019 Apr 29. PMID 31037340